CLINICAL TRIAL: NCT02275676
Title: Influence of Disease Activity of Inflammatory Bowel Disease on Resting Energy Expenditure and Nutritional Status
Brief Title: Resting Energy Expenditure and Nutritional Status in IBD
Acronym: CEDERN-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Dr. med. Hauke Heinzow, Doktor, University Hospital Muenster
Other Study IDs: CEDERN1
Record Dates: First submitted 2014-10-13; First posted 2014-10-27 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Inflammatory Bowel Disease; Malnutrition
Keywords: Inflammatory bowel disease; Nutritional Status; Malnutrition; Resting Energy Expenditure
MeSH Terms: conditions — Inflammatory Bowel Diseases; Malnutrition | interventions — Calorimetry, Indirect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Inflammatory bowel disease: Patients with active and inactive inflammatory bowel disease
  Interventions: Other: bioelectrical impedance analysis; Other: indirect calorimetry

INTERVENTIONS:
Other: bioelectrical impedance analysis
Other: indirect calorimetry

SUMMARY:
Nutrient deficiencies occur frequently in IBD patients. The absorption rate of nutrients in IBD is often limited by chronic inflammation, but is also commonly reduced by missing intestinal segments due to previous operations. Patients are predominantly affected by malnutrition, which is often resembled by weight loss, specific micronutrient deficits such as iron deficiency, vitamin B12 deficiency, folic acid deficiency, vitamin D deficiency and zinc depletion. The etiology of nutritional problems is multifactorial and not exclusively limited to active phases of the disease. Causes of malnutrition can be inadequate food intake, maldigestion, malabsorption or increased nutritional requirement. Malnutrition itself is associated with a delayed recovery of impaired wound healing, reduced quality of life and longer hospital stays. Therefore, observation and modification of the nutritional status should be an integral part of therapy in IBD patients.

The primary objective of our study is to investigate the influence of the disease on the resting energy expenditure and nutritional status during acute inflammation and clinical remission of the disease. Secondary objectives are to assess possible nutritional deficiencies. On the other hand it is well known that patients with IBD are at increased risk for coronary heart disease. Therefore, another secondary focus of our observational study is whether the composition of the HDL proteins is changed towards pro-atherogenic HDL-proteins and whether possible changes occur in patients in clinical remission or with active disease.

DETAILED DESCRIPTION:
Primary objective of the study is to investigate the influence of the disease activity on the resting energy expenditure and the nutritional status in patients with chronic inflammatory bowel disease (IBD). The impact of IBD on the nutritional status and the resting energy expenditure is currently not fully understood. IBD includes two different disease entities, Crohn's disease and ulcerative colitis. Both are characterized by diarrhea, loss of weight, rectal bleeding and abdominal discomfort (abdominal pain, flatulence). In patients with IBD malabsorption, one-sided nutritional behavior, food abandonment, malnutrition, nutrient deficiency and weight loss are common issues. Malnutrition is associated with delayed recovery, impaired wound healing, reduced quality of life and prolonged hospital stay. The malnutrition is not limited to active disease state. Rates for malnutrition in patients with Crohn's disease range from 20 - 85%. Hence, the assessment of the nutritional status is important in the treatment of patients with IBD. Different methods are used to assess the impact of the disease activity on the nutritional status. To investigate the resting energy expenditure the well evaluated indirect calorimetry is used. The principle of the measurement is based on determination of the oxygen absorption during inspiration and the simultaneous determination of the release of carbon dioxide during expiration. The use of bioelectrical impedance analysis (BIA) is a widespread measurement to assess the composition of the body. BIA allows the determination of the fat-free mass, total body water, body cell mass, fat mass and extracellular mass.

Both measurements are non-invasive and reproducible. Additionally different blood parameters are determined such as HDL-subgroups, vitamin b12, folic acid, vitamin K, vitamin D, 25-hydroxy-vitamin D3, zinc, ferritin, albumin, citrulline and routine laboratory (blood count, serum chemistry, coagulation) . Moreover the quality of life is measured through a suitable questionnaire (Gastrointestinal Life Quality Index) as well as the subjective global assessment to estimate the nutritional status.

Furthermore, a secondary aim of the study is to investigate the correlation of HDL-subgroups and the severity of the IBD activity. High-Density-Lipoproteins are a heterogeneous group of lipoproteins with both anti-atherogenic and multiple anti-inflammatory properties. Recent research showed that the quality of HDL-particle is even more important than the quantity. It could be shown that changes in the composition of the HDL could cause an inflammatory status and thus affect the activity of chronic inflammatory disease. Therefore, it is the aim of the study to investigate if changes in the composition of HDL-proteins towards pro-atherogenic HDL-proteins exist.

The study will take place at the University Hospital of Muenster, Germany. Patients who are suitable for participating in the study will be measured and counseled during their regular out-clinic visits. Each patient has to undergo the procedure while they are in an active state of the disease and during remission. It is expected to include 200 patients over 2 years.

ELIGIBILITY:
Inclusion Criteria:

* inflammatory bowel disease
* male and female between 18-80 years
* patient fully able to understand the study concept and to give his or her written consent

Exclusion Criteria:

* underlying malignant disease
* Diabetes mellitus, Type I or II
* Pregnancy
* Lactating
* chronic alcohol or drug abuse
* known anorexia nervosa or binge eating disorder
* known metabolic disorders, such as e.g. Cushing disease, hypothyroidism
* Participation in other interventional studies within the last 6 months prior to study enrollment
* patient not fully able to understand the study concept and to give his or her written consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with active or inactive inflammatory bowel disease at our medical tertiary referral center, Muenster Germany
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
change in bioelectrical impedance analysis (BIA) | change from baseline in BIA at 6 month and at 12 month
  e.g. fat free mass, total body water, body cell mass
Change in resting energy expenditure (REE) | change from baseline in REE at 6 month and at 12 month
  Resting energy expenditure measured by indirect calorimetry (kcal per day)

SECONDARY OUTCOMES:
change in HDL subgroup analysis | day 1, every 6 month up to 12 month
change in plasma citrulline level | day 1, every 6 month up to 12 month
change in plasma vitamine levels and plasma zinc level | day 1, every 6 month up to 12 month
  Vitamin B12, Vitamin K, Vitamin D

OTHER OUTCOMES:
change in fecal Calprotectin level | day 1, every 6 month up to 12 month
change in live quality questionnaire | day 1, every 6 month up to 12 month
  Gastrointestinal Quality of Life Index by Eypasch

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lenze, Dr., Principal Investigator — University Hospital Muenster, Germany; Hauke Heinzow, Dr., Principal Investigator — University Hospital Muenster, Germany
Locations (1):
- University Hospital Muenster, Münster, Germany